CLINICAL TRIAL: NCT01366833
Title: Management of Malignant Dysphagia: Stent vs. Stent Plus Endoluminal Brachytherapy for the Palliation of Dysphagia in Metastatic Esophageal Cancer
Brief Title: Optimal Management of Malignant Dysphagia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Lorenzo Ferri, Dr., McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MalignantDysphagia
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Malignant Dysphagia; Esophageal Cancer
Keywords: Dysphagia; Esophagus; Cancer; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders; Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-expanding stent alone (Active Comparator): All patients in Arm A will receive self-expanding stent alone
  Interventions: Procedure: Stent insertion
- Brachytherapy and Stent therapy (Experimental)
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — Patients in arm B will receive a single dose of brachytherapy (10Gy) via a 10 or 13 mm catheter within 10days of stent insertion. Patients on the study will not be given preferential treatment, and will not be prioritized over patients treated with brachytherapy not on the study.
  Arms: Brachytherapy and Stent therapy
Procedure: Stent insertion — After placement of clips to mark the proximal and distal extent of the tumor, an endoscopically placed self-expanding metallic stent (WallFlex™ Partially Covered Esophageal Stent by Boston Scientific) will be inserted within 10 days of recruitment. This will be the only intervention in Arm A patients.
  Arms: Self-expanding stent alone

SUMMARY:
According to the Canadian Cancer Society there are approximately 1700 new cases of esophageal cancer per year in Canada. As most of these patients are diagnosed in advanced stages of the disease, 1800 deaths are estimated from this cancer annually . Progressive dysphagia is the most common presenting symptom and impacts not only the patient's quality of life but the ability to tolerate life prolonging treatments such as systemic chemotherapy.

Although there are several therapeutic modalities to alleviate malignant dysphagia including laser, photodynamic therapy and cryotherapy , the use of stents and radiotherapy are the most commonly employed. However, the optimal approach to effective, timely treatment of malignant dysphagia remains a challenge. The investigators conducted a preliminary retrospective review to investigate such palliation procedures and found that a multi-modality approach may yield the most favourable results .

Therefore, our clinical trial will examine the effectiveness of adding a single dose of brachytherapy to patients with severe dysphagia who have already been treated with a endoscopically placed self-expanding metallic stent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed esophageal/gastroesophageal (GEJ) cancer (Siewert Type I and Type II only) of any histology on biopsy
* Dysphagia score ≥2
* Stage IV cancer/Metastatic disease

Exclusion Criteria:

* Expected life expectancy < 3 months
* Inability to undergo stent insertion
* Siewert Type III gastroesophageal cancer
* Esophageal-Airway fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To investigate the change in dysphagia score (0-4 Likert scale) measured at baseline and at 10 weeks | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ferri, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Monisha Sudarshan, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Marc David, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; David Roberge, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Serge Mayrand, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Kevin Waschke, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Eleanor Eckert, Nutritionist, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Myriam Martel, RN, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada